CLINICAL TRIAL: NCT03302377
Title: Fit for Two: Feasibility and Acceptability of Incorporating Wearable Trackers Into Clinical Care for Pregnant Women With Diabetes
Brief Title: Fit for Two: Incorporating Wearable Trackers Into Clinical Care for Pregnant Women With Diabetes (FFT)
Acronym: FFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Britta Larsen, Assistant Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CFM281R
Record Dates: First submitted 2017-09-29; First posted 2017-10-05 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Physical Activity; Type 2 Diabetes Mellitus
Keywords: Feasibility
MeSH Terms: conditions — Motor Activity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: As this is a feasibility study, all participants will receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity intervention (Experimental): Participants will receive an individual counseling session in the clinic to help them set physical activity and step goals. They will then receive a Fitbit wrist monitor and help personalizing the Fitbit app. They will send weekly emails to their physicians reporting their goals and current activity. They will return at 12 weeks to engage in a semi-structured interview to give their overall impressions of the intervention.
  Interventions: Behavioral: physical activity counseling & Fitbit

INTERVENTIONS:
Behavioral: physical activity counseling & Fitbit — Participants will receive individual counseling & guidance in goal setting, then will receive a Fitbit wrist monitor and guidance in personalizing the Fitbit features

SUMMARY:
This study will investigate the feasibility of an intervention to increase physical activity in pregnant women with diabetes by incorporating a brief in-person counseling session and Fitbit activity trackers into routine clinical care

DETAILED DESCRIPTION:
This is a small, one-armed pilot study testing a physical activity intervention for pregnant patients with diabetes. The intervention will use both counseling and technology (a FitBit physical activity tracker and smartphone app) to create an individualized, interactive program for each patient. The primary aims of the study are to assess the feasibility of recruiting patients and implementing the program in the clinical setting, and the acceptability of the program for patients and clinicians. Participants will receive a counseling session based on the principles of motivational interviewing to help them set physical activity and step goals, then the interventionist will help them personalize the Fitbit app to their goals. Participants are instructed to continue adaptive goal setting and email their goals and activity weekly to their physicians. In addition to assessing feasibility and acceptability, we will also evaluate change in activity to explore potential efficacy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes or gestational diabetes
* currently pregnant
* in week 5-25 of gestation
* under active (<100 minutes/week of physical activity)
* access to a smartphone

Exclusion Criteria:

* any medical condition that would make unsupervised activity unsafe or unfeasible, as determined by their physician
* moving from the area within 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for pregnant patients, so all participants will be female
Enrollment: 19 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Retention | 12 weeks
  Determined by retention (%)
Acceptability | 12 weeks
  Determined by participant feedback (% indicating satisfaction with intervention)
Feasibility of recruitment | baseline
  Determined by percent of those screened who enroll in the study

SECONDARY OUTCOMES:
Physical activity change | 12 weeks
  Change in objectively measured physical activity from baseline to follow-up as measured by hip-worn ActiGraph GT3X+ accelerometers, adjusting for baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers

REFERENCES:
- [Derived] Larsen B, Micucci S, Hartman SJ, Ramos G. Feasibility and Acceptability of a Counseling- and mHealth-Based Physical Activity Intervention for Pregnant Women With Diabetes: The Fit for Two Pilot Study. JMIR Mhealth Uhealth. 2020 Oct 21;8(10):e18915. doi: 10.2196/18915. PMID 33084584